CLINICAL TRIAL: NCT06427694
Title: The Low-Dose Interleukin-2 For The Reduction Of Vascular Inflammation In Acute Coronary Syndromes -Clinical Outcomes And Follow-up Study
Brief Title: Low-Dose IL-2 For The Reduction Of Vascular Inflammation In ACS -Clinical Outcomes & Follow-up Study
Acronym: IVORY-FINALE
Status: Recruiting | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Joseph Cheriyan, MBChB, MA, FRCP, FESC, FACC, Dr Joseph Cheriyan, Consultant Clinical Pharmacologist/Affilitated Associate Professor, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: IVORY-FINALE (A096877); 339102 (Other: IRAS)
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — aldesleukin; Glucose; Water

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aldesleukin: Aldesleukin loading dose 1.5 x 10^6 IU followed by maintenance dose of 1.5 x 10^6 IU
  Interventions: Drug: Aldesleukin
- Placebo: Dextrose 5%
  Interventions: Drug: Dextrose 5% in water

INTERVENTIONS:
Drug: Aldesleukin — IL2 antagonist
  Other Names: Proleukin
  Groups: Aldesleukin
Drug: Dextrose 5% in water — matched placebo to active
  Other Names: Dextrose
  Groups: Placebo

SUMMARY:
The preceding IVORY trial (NCT04241601) has completed. As atherosclerosis and its complications are driven by inflammation the investigators hypothesise that treatment with low-dose IL2 may reduce adverse cardiovascular outcomes compared to placebo.

In this follow-up study, the investigators aim to collect cardiovascular clinical outcome data for patients who completed the IVORY clinical trial and will look at major adverse cardiovascular events (MACE), defined as cardiovascular death, non-fatal myocardial infarction, resuscitated cardiac arrest, ischaemic stroke, or unplanned coronary revascularization. In addition, data on adverse events such as all cause death, haemorrhagic stroke, new atrial fibrillation, ventricular arrhythmias, hospitalisation due to cardiovascular causes (e.g. stable and unstable angina, TIAs, heart failure), amputations and revascularisation due to peripheral vascular disease.

DETAILED DESCRIPTION:
A heart attack occurs when there is reduced blood flow to heart muscle cells which results from narrowings or blockages in walls of blood vessels supplying the heart, due to fatty deposits and inflammatory cells that build up over time. This build-up leads to heart muscle damage called a heart attack.

The immune system plays an important role in both the development of the narrowings and the damage to the heart muscle during a heart attack. Studies have shown that there is a lower level of protective immune cells called regulatory T-cells (Tregs) in heart attack patients. Increasing the number of circulating Tregs may have a direct effect in reducing the inflammation in arteries, preventing further narrowings in blood vessels and improving heart muscle function. Aldesleukin, also known as interleukin-2 (IL2), is a medicine that stimulates the production of Treg cells when given at low doses. The effectiveness of IL2 in influencing the immune system was tested in a phase 2 trial, IVORY.

Participants were recruited to the IVORY trial following a sudden narrowing/blockages in walls of blood vessels to the heart resulting in a heart attack (Acute Coronary Syndrome (ACS)). Participants were randomised to receive either low dose IL2 or placebo, researchers and participants were blinded to the treatment allocation. Participants underwent two PET/CT (Positron emission tomography-computed tomography) scans to observe change of inflammation in the blood vessels from baseline between the two trial groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants who completed the full per-protocol treatment regime of low-dose IL2 or placebo having attended the final dosing visit in the IVORY trial. IVORY patients who previously consented to have their medical records inspected in the IVORY trial and who have already passed away at the commencement of IVORY-FINALE will also be included in analyses

Exclusion Criteria:

* Patients who decline participation
* Patients who did not consent to being contacted about future research
* Patients who were withdrawn from the IVORY trial for any reason

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of the IVORY trial (NCT04241601) and who consented to be contacted for future research received all scheduled doses of either placebo or IL2 and are alive at the time of data collection will be approached.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2030-02-11 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular outcomes | 1 year from when initially dosed in preceding IVORY trial
  Number of major adverse cardiovascular outcomes
Major adverse cardiovascular outcomes | 2 years from when initially dosed in preceding IVORY trial
  Number of major adverse cardiovascular outcomes
Major adverse cardiovascular outcomes | 5 years from when initially dosed in preceding IVORY trial
  Number of major adverse cardiovascular outcomes

SECONDARY OUTCOMES:
Death due to cardiovascular causes | 1 year from when initially dosed in preceding IVORY trial
  Number of deaths due to cardiovascular causes comparing IL2 to placebo
Deaths due to cardiovascular causes comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Number of deaths due to cardiovascular causes comparing IL2 to placebo
Deaths due to cardiovascular causes comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Number of deaths due to cardiovascular causes comparing IL2 to placebo
Resuscitated cardiac arrests comparing IL2 to placebo | 1 year from when initially dosed in preceding IVORY trial
  Numbers of resuscitated cardiac arrests comparing IL2 to placebo
Resuscitated cardiac arrests comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Numbers of resuscitated cardiac arrests comparing IL2 to placebo
Resuscitated cardiac arrests comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Numbers of resuscitated cardiac arrests comparing IL2 to placebo
Non-fatal MI (including NSTEMI and STEMI) comparing IL2 to placebo | 1 year from when initially dosed in preceding IVORY trial
  Number of non-fatal MI (including NSTEMI and STEMI) comparing IL2 to placebo
Non-fatal MI (including NSTEMI and STEMI) comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Number of non-fatal MI (including NSTEMI and STEMI) comparing IL2 to placebo
Non-fatal MI (including NSTEMI and STEMI) comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Number of non-fatal MI (including NSTEMI and STEMI) comparing IL2 to placebo
Ischaemic strokes comparing IL2 to placebo | 1 year from when initially dosed in preceding IVORY trial
  Number of ischaemic strokes comparing IL2 to placebo
Ischaemic strokes comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Number of ischaemic strokes comparing IL2 to placebo
Ischaemic strokes comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Number of ischaemic strokes comparing IL2 to placebo
Unplanned coronary vascularisations comparing IL2 to placebo | 1 year from when initially dosed in preceding IVORY trial
  Number of unplanned coronary vascularisations comparing IL2 to placebo
Unplanned coronary vascularisations comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Number of unplanned coronary vascularisations comparing IL2 to placebo
Unplanned coronary vascularisations comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Number of unplanned coronary vascularisations comparing IL2 to placebo
Hospitalisations due to cardiovascular causes comparing IL2 to placebo | 1 year from when initially dosed in preceding IVORY trial
  Number of hospitalisations due to cardiovascular causes comparing IL2 to placebo
Hospitalisations due to cardiovascular causes comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Number of hospitalisations due to cardiovascular causes comparing IL2 to placebo
Hospitalisations due to cardiovascular causes comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Number of hospitalisations due to cardiovascular causes comparing IL2 to placebo
All-cause deaths comparing IL2 to placebo | 1 year from when initially dosed in preceding IVORY trial
  Number of all-cause deaths comparing IL2 to placebo
All-cause death comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Number of all-cause deaths comparing IL2 to placebo
All-cause death comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Number of all-cause deaths comparing IL2 to placebo
Hospitalisations due to symptoms from heart failure (incl admission due to pulmonary oedema and congestive heart failure) comparing IL2 to placebo | 1 year from when initially dosed in preceding IVORY trial
  Number of hospitalisations due to symptoms from heart failure (incl admission due to pulmonary oedema and congestive heart failure) comparing IL2 to placebo
Hospitalisations due to symptoms from heart failure (incl admission due to pulmonary oedema and congestive heart failure) comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Number of hospitalisations due to symptoms from heart failure (incl admission due to pulmonary oedema and congestive heart failure)comparing IL2 to placebo
Hospitalisations due to symptoms from heart failure (incl admission due to pulmonary oedema and congestive heart failure) comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Number of hospitalisation due to symptoms from heart failure (incl admission due to pulmonary oedema and congestive heart failure) comparing IL2 to placebo
Revascularisations for peripheral vascular disease comparing IL2 to placebo | 1 year from when initially dosed in preceding IVORY trial
  Number of revascularisations for peripheral vascular disease comparing IL2 to placebo
Revascularisations for peripheral vascular disease comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Number of revascularisations for peripheral vascular diseasecomparing IL2 to placebo
Revascularisations for peripheral vascular disease comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Number of revascularisations for peripheral vascular disease comparing IL2 to placebo
Amputations due to peripheral vascular disease comparing IL2 to placebo | 1 year from when initially dosed in preceding IVORY trial
  Number of amputations due to peripheral vascular disease comparing IL2 to placebo
Amputations due to peripheral vascular disease comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Number of amputations due to peripheral vascular disease comparing IL2 to placebo
Amputations due to peripheral vascular disease comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Number of amputations due to peripheral vascular disease comparing IL2 to placebo
Haemorrhagic strokes comparing IL2 to placebo | 1 year from when initially dosed in preceding IVORY trial
  Number of haemorrhagic strokes comparing IL2 to placebo
Haemorrhagic strokes comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Number of haemorrhagic strokes comparing IL2 to placebo
Haemorrhagic strokes comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Number of haemorrhagic strokes comparing IL2 to placebo
New atrial fibrillation diagnosis comparing IL2 to placebo | 1 year from when initially dosed in preceding IVORY trial
  Number of new atrial fibrillation diagnoses comparing IL2 to placebo
New atrial fibrillation diagnosis comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Number of new atrial fibrillation diagnoses comparing IL2 to placebo
New atrial fibrillation diagnosis comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Number of new atrial fibrillation diagnoses comparing IL2 to placebo
Ventricular arrhythmia (sustained ventricular tachycardia and ventricular fibrillation) comparing IL2 to placebo | 1 year from when initially dosed in preceding IVORY trial
  Number of ventricular arrhythmia episodes (sustained ventricular tachycardia and ventricular fibrillation) comparing IL2 to placebo
Ventricular arrhythmia (sustained ventricular tachycardia and ventricular fibrillation) comparing IL2 to placebo | 2 years from when initially dosed in preceding IVORY trial
  Number of ventricular arrhythmia episodes (sustained ventricular tachycardia and ventricular fibrillation) comparing IL2 to placebo
Ventricular arrhythmia (sustained ventricular tachycardia and ventricular fibrillation) comparing IL2 to placebo | 5 years from when initially dosed in preceding IVORY trial
  Number of ventricular arrhythmia episodes (sustained ventricular tachycardia and ventricular fibrillation) comparing IL2 to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MBChB, FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
On completion of the study the data will be analysed and tabulated and a Final Study Report prepared. Data will be published in an open access journal.